CLINICAL TRIAL: NCT06427824
Title: Comprehensive Geriatric Assessment Utilization for Bladder Cancer Patients Undergoing Radical Cystectomy: A Randomized Controlled Trial
Brief Title: Comprehensive Geriatric Assessment (Tests) for Bladder Cancer Participants Undergoing Radical Cystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB23-0773
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer
Keywords: cystectomy; radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Surgical Procedures, Operative; Patient Discharge; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants Who Watch Educational Videos Before Surgery (Experimental): Participants in this group will attend an educational session in a conference room that includes 4 learning modules on strategies to reduce mobility loss, improve medication management, prevent delirium, and to document what matters most before and after surgery (cystectomy). These learning modules will be in video format. Participants will watch videos to learn about pre/post surgical strategies and they will receive informational handouts after watching the videos. The study team will also ask participants to fill out questionnaires/surveys before and after surgery.
  Interventions: Other: Educational Video Modules on Risk Prevention Before and After Cystectomy (Surgery); Other: Questionnaires
- Participants Who Watch Educational Videos Before Surgery and Receive Geriatric Follow Up Services (Experimental): Participants in this group will also attend an educational session in a conference room that includes 4 learning modules on strategies to reduce mobility loss, improve medication management, prevent delirium, and to document what matters most before and after surgery (cystectomy). These learning modules will be in video format. Participants will watch videos to learn about pre/post surgical strategies and they will receive informational handouts after watching the videos. The study team will also ask participants to fill out questionnaires/surveys before surgery.
  In addition to attending the educational program (via video) and receiving informational handouts, participants in this group will also meet with the study doctor and/or members of the study team after surgery to help plan their hospital discharge and reinforce/use the strategies they learned in the educational session after surgery.
  Interventions: Other: Educational Video Modules on Risk Prevention Before and After Cystectomy (Surgery); Other: Geriatric Service/ Discharge Planning; Other: Questionnaires

INTERVENTIONS:
Other: Educational Video Modules on Risk Prevention Before and After Cystectomy (Surgery) — An educational program designed by geriatricians, surgeons, anesthesiologists and palliative care physicians to help people with bladder cancer who plan to receive a cystectomy learn strategies to improve their mobility, medication management, mental clarity/delirium and how they document important side effects or health issues after surgery.
Other: Geriatric Service/ Discharge Planning — A geriatric team will meet with participants after surgery to help them reinforce the strategies they learned in the education video sessions. As part of a geriatric service, this team will also help participants plan/coordinate their discharge from the hospital after surgery.
  Arms: Participants Who Watch Educational Videos Before Surgery and Receive Geriatric Follow Up Services
Other: Questionnaires — These questionnaires will ask about the participants' mobility, frailty, quality of life and additional health/risk factors before and after surgery.

SUMMARY:
This study focuses on providing an educational program for people/participants with bladder cancer who plan to have a cystectomy (surgery) as part of their standard care. Participants in this study will watch videos designed to teach them strategies to help lower their risk of experiencing negative side effects (such as mobility problems, issues with taking medication, and poor quality of life) before and after they have surgery. They will also be asked to fill out questionnaires.

DETAILED DESCRIPTION:
This study focuses on providing an educational program for participants/people with bladder cancer who plan to have a cystectomy (surgery) as part of their standard care. Participants in this study will watch videos designed to teach them strategies to help lower their risk of experiencing negative side effects (such as mobility problems, issues with taking medication, and poor quality of life) before and after they have surgery. The goal of this study is to educate people with bladder cancer and ask them to also fill out questionnaires about the education program and if they used any of the strategies that learn during the study.

Participants in this study will be divided into two different study groups (one group that watches educational videos before surgery and one group that watches educational videos before surgery and also receives geriatric services and follow up visits after surgery). Each participant will be randomized (randomly assigned) to one of two study groups. That means that there is a 50/50 chance (like flipping a coin) that each participant will end up in either group.

ELIGIBILITY:
Inclusion Criteria

* Participants capable of giving consent
* Participants undergoing radical cystectomy (both for curative and palliative intent) for bladder cancer diagnosed by tissue pathology with urinary diversion at the University of Chicago
* Participants undergoing neoadjuvant chemotherapy will be included
* Participants will be included regardless of gender, race or ethnicity
* Participants greater than or equal to 65 years of age

Exclusion Criteria

* Radical cystectomy for non-oncologic indications
* Palliative cystectomy for cancers other than bladder cancer (i.e. prostate, rectal, cervical)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Referred to Educational Program | 90 days
  Assess the feasibility of an educational program designed for participants undergoing radical cystectomy by measuring the number of participants referred to the study team/program.

SECONDARY OUTCOMES:
Survey responses from participants who completed some or all of educational program | 90 days
  Assess the acceptability of an educational program designed for participants undergoing radical cystectomy by measuring/surveying the number of study participants who completed at least some of the intervention.
Number of self-reported interventions/strategies used among participants after watching educational videos | 90 days
  Assess the adoptability of an educational program designed for participants undergoing radical cystectomy by measuring the number of self-reported interventions that participants reported after the educational program
30-day Hospital Readmission Rates Among All Participants | 30 days
  Assess impact of educational program by comparing the differences between hospital readmission rate at 30 days between both study cohorts.
90-day Hospital Readmission Rates Among All Participants | 90 days
  Assess impact of educational program by comparing the differences between hospital readmission rate at 90 days between both study cohorts.
Complication Rates Reported Among Participants | 90 days
  Assess impact of educational program by comparing the differences between complication rates reported among study participants in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Piyush Agarwal, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF